CLINICAL TRIAL: NCT05520801
Title: The Treatment and Prognosis of Primary Hepatobiliary Cancer: A Cohort Study in Central China
Brief Title: Primary Hepatobiliary Cancer Cohort of Central China
Acronym: CCGLC-002
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Chinese Cooperative Group of Liver Cancer (Other); Chen Xiao-ping Foundation for the Development of Science and Technology of Hubei Province (Other); Haplox Biotechnology Co., Ltd. (Industry); Geneplus-Beijing Co. Ltd. (Industry); YuceBio Technology (Unknown); Gelesis, Inc. (Industry)
Responsible Party: Principal Investigator, Zhang Bi Xiang, MD, Chairman of Department of General Surgery, Tongji Hospital
Other Study IDs: TJ-IRB20210935
Record Dates: First submitted 2022-01-23; First posted 2022-08-30 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Hepatocellular Carcinoma; Biliary Tract Neoplasms
Keywords: Primary Hepatobiliary Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tissue, blood, urine, feces, ascites, bile samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry is designed as a longitudinal cohort study of patients diagnosed with primary hepatobiliary cancer in Tongji Hospital, Wuhan. This study collects the clinical-pathological features of hepatic malignant tumors and the current status of patients who received comprehensive treatment based on surgical treatment since 1998.

DETAILED DESCRIPTION:
This longitudinal observational cohort study was designed to make standardized settlements, statistical treatments, and comprehensive analysis of primary hepatobiliary cancers in middle China, which summarize and estimate the population, tumor staging, treatment mode, clinical-pathological characteristics, and the prognosis, to provide evidence for standardized treatment of hepatobiliary cancers.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old,
2. life expectancy is at least 6 months.
3. Diagnosed as primary liver cancer or biliary malignant tumor by histopathology or confirmed by imaging as HCC (by the AASLD or guidance for the diagnosis and treatment of primary liver cancer of China (version 2022).
4. At least one measurable lesion (RECIST v1.1)
5. Subjects volunteer to participate in the study and sign informed consent.

Exclusion Criteria:

Patients with one or more of the following criteria should be excluded:

1. CT or MRI shows no measurable lesions (RECIST v1.1).
2. Patients after comprehensive assessment are considered by the investigators to be unsuitable for participating in the study.
3. Incomplete baseline or follow-up data
4. Suffering from more than two kinds of primary tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed as primary hepatobiliary cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From diagnosis or treatment initiation to date of death due to any cause, or last known vital status date, up to 2 years
  Time of death will be obtained by telephone interview or medical treatment records.
Progression-free survival (PFS) | From treatment initiation for advanced or metastatic HCC to the first date of disease progression for any cause up to 2 years
  Patients lost for follow up or withdrawn from the study will be censored at the last disease assessment date
Disease Control Rate (DCR) | From treatment initiation to SD, CR or PR, up to 2 years
  The proportion of patients who had either stable disease (SD) for ≥ 6 months, a CR or PR after initiation of treatment for HCC
Duration of Response (DOR) | From treatment initiation to PD, up to 2 years
  DOR is the duration from the first assessment of the tumor was CR or PR to the time that the first assessment for PD or date of death from any cause
Objective response rates (ORR) | From treatment initiation to CR or PR, up to 2 years
  Percentage of patients whose tumors have a complete or partial response to treatment.

SECONDARY OUTCOMES:
Time of recurrence | From date of diagnosis until the date of cancer recurrence or date of death from any cause, whichever came first, assessed up to 10 years
  Time of recurrence will be obtained by telephone interview or medical treatment records
Time of metastasis | From date of diagnosis until the date of cancer metastasis or date of death from any cause, whichever came first, assessed up to 10 years
  Time of metastasis will be obtained by telephone interview or medical treatment records
Quality of Life (QoL) after treatment | From date of diagnosis until the date of cancer recurrence or date of death from any cause, whichever came first, assessed up to 10 years
  Life quality of every subject will be assessed every 3 months according to the FACT-Hep questionnaire, which assesses generic HRQL concerns and disease-specific issues.

CONTACTS AND LOCATIONS:
Overall Officials: Bixiang Zhang, Study Chair — Tongji Hospital; Zeyang Ding, Principal Investigator — Tongji Hospital
Locations (1):
- Hepatic Surgery Center, Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China